CLINICAL TRIAL: NCT05090085
Title: Clinical Assessment of Dimethyl Sulfoxide in OT Primer Prior to Dental Adhesive: Randomized Controlled Trial
Brief Title: Invivo Clinical Assessment of Dimethyl Sulfoxide in OT Primer Prior to Dental Adhesive
Acronym: DMSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Horus University (Other)
Responsible Party: Principal Investigator, Omar Abdelaziz Ismail, Principal Investigator, BDS, MSc, FINDOS Candidate Cariology and Restorative Dentistry. Member of the Adhesive group of Turku. Finland, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTurku Clinical DMSO
Record Dates: First submitted 2021-10-09; First posted 2021-10-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-02

CONDITIONS: Dental Diseases
Keywords: DMSO
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In our clinical trial, double blinding will be performed, the participants and assessors will be blinded to the type of material used to reduce performance and ascertainment bias and also reduce biased estimates of treatment effects. The operator cannot be blinded in this trial because of the difference in the application procedures of each restorative material. Therefore, the operator (O.I.) will take care to treat the two allocation groups as equally as possible by standardizing the care of participants, frequency of follow-ups and management of complications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3M Adper Single Bond2 (Active Comparator): O.I. will clean the labial surface of the tooth with polishing paste and brush Roughening of the surface may be needed by the diamond point The tooth will be isolated by a rubber dam. Apply etchant for 30 s for enamel and 15 s for dentin. Rinse thoroughly with water for 15 s. blot-drying with paper tissue was carefully performed leaving the dentin surface slightly moist. Active application of consecutive coats of the adhesive for 15 s. Gently air for 5 s. Light cure for 10 s. Composite build ups (Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA) were performed in increments and individually light-cured for 20 s. Light curing of all resin materials was performed using (3M Elipar Curing Light) delivering 1100 mW/cm2.
  Interventions: Other: 3M Adper Single Bond2; Other: Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA); Other: 3m ESPE etch
- DMSO application before 3M Adper Single Bond2, etch and rinse adhesive (Experimental): The same steps of the comparator group with an additional step, after dentin etching and humidity control, dentin pretreatments were performed consisting of active application of 10% DMSO/H2O (OT Primer, OT Dent) solutions on etched-dentin for 1 minute followed by 20 seconds of air drying then apply adhesive.
  Interventions: Other: 3M Adper Single Bond2; Other: Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA); Other: 3m ESPE etch; Other: OT Primer

INTERVENTIONS:
Other: 3M Adper Single Bond2 — Two-step etch and rinse dental adhesive system
Other: Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA) — Composite Resin
Other: 3m ESPE etch — 32% phosphoric acid
Other: OT Primer — Dimethyl Sulfoxide DMSO [(CH3)2SO] is a polar aprotic solvent that dissolves both polar and non-polar compounds.
  Other Names: 10% DMSO/H2O
  Arms: DMSO application before 3M Adper Single Bond2, etch and rinse adhesive

SUMMARY:
This study is conducted to assess the clinical effectiveness of 10% Dimethyl Sulfoxide in OT Primer prior to two step etch and rinse dental adhesive on the durability of composite restoration.

DETAILED DESCRIPTION:
Randomized Controlled Clinical Trial After the power analysis calculation, 74 cervical lesions will be included in this study. Half of them will be pretreated with 10% DMSO/H2O (Dimethyl Sulfoxide/Water, OT Primer, OT Dent). Control groups will be bonded with SB (Single Bond2, 3M ESPE). Cavities will be restored with nanohybrid composite restoration (Z350 XT, 3M ESPE) under rubber dam isolation. Follow-ups will be performed by double-blinded evaluators at baseline and after 6m, 12m, 24m, and 36m using the FDI criteria. Photographic documentation will be performed for all restorations.

Sample size calculation The sample size was calculated based on a previous study by Vural et al in 2020, in which success rate of resin composite cervical restorations was 73% after 36 months. By implementing a two tailed Z test for difference between two independent proportions with an alpha level of 5% and a power of 80%. The minimum sample size needed was 30 per group in order to detect a difference of 25%. Sample size was increased by 25% to compensate for possible dropouts to reach 37 teeth per group. Sample size was performed using G*Power version 3.1.9.2 for windows.

Statistical Analyses Data was analyzed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium). Categorical data was described as frequency and percentage, intergroup comparisons between interventions was performed using Chi-Square test with statistical significance level set at (P ≤ 0.05), intragroup comparison within each intervention was performed using the Cochran's Q test with statistical significance level set at (P ≤ 0.0083) after Bonferroni correction. Relative risk was used to assess the clinical significance. Survival rate was analyzed using Kaplan-meier and Log-rank test. The confidence limit was set at 95% with 80% power and all tests were two tailed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Carious Cervical Lesions (CCL).
* Co-operative patients approved to participate in the study.
* Pulp is asymptomatic vital teeth.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Patients with Non-Carious Cervical Lesions (NCCL).
* Xerostomia
* Bruxism and visible wear facets in the posterior dentition.
* Known inability to return for recall appointments.
* Fractured or visibly cracked candidate tooth.
* Current desensitizing therapy, including desensitizing dentifrices or other over-the-counter (OTC) products.
* Long-term use of anti-inflammatory, analgesic, or psychotropic drugs.
* Pregnancy or breast-feeding (potential conflicts with recall dates.
* Allergies to ingredients of resin-based restorative materials.
* Orthodontic appliance treatment within the previous three months.
* Abutment teeth for fixed or removable prostheses.
* Teeth or supporting structures with any symptomatic pathology.
* Existing periodontal disease or periodontal surgery within the previous three months.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Functional (Number of Restorations with change of marginal adaptation) | [Time Frame: Day 0, Month 12, Month 24, Month 36]
  FDI criteria for evaluation of restorations, percentage score.
  * Score: Properties.
  * Clinically excellent/ very good: Harmonious outline, no gaps, no white or discolored lines.
  * Clinically good: Marginal gap (<150 μm), White lines. Or Small marginal fracture removable by polishing. or Slight ditching, slight step/flashes, minor Irregularities.
  * Clinically sufficient/satisfactory: Gap < 250 μm not removable. Or Several small marginal fractures. Or Major irregularities, ditching or flash, steps.
  * Clinically unsatisfactory: Gap > 250 μm or dentine/base exposed. Or Severe ditching or marginal fractures. or Larger irregularities or steps (repair necessary).
  * Clinically poor: Restoration (complete or partial) is loose but in situ. Or Generalized major gaps or irregularities.

SECONDARY OUTCOMES:
Esthetic (Number of Restorations with change of color match and translucency) | [Time Frame: Day 0, Month 12, Month 24, Month 36]
  FDI criteria for evaluation of restorations, percentage score.
  * Score: Properties
  * Clinically excellent/ very good: Good color match, no difference in shade and/or translucency.
  * Clinically good: Minor deviations in shade and/or translucency.
  * Clinically sufficient/satisfactory: Distinct deviation but acceptable. Does not affect esthetics: 1. more opaque ,2.
  more translucent ,3. darker,4. brighter.
  * Clinically unsatisfactory: Localized clinically deviation that can be corrected by repair: 1.Too opaque, 2.Too translucent,3. Too dark, 4.Too bright.
  * Clinically poor: Unacceptable. Replacement necessary.
Biological (Number of Restorations with change of caries adjacent to the restoration) | [Time Frame: Day 0, Month 12, Month 24, Month 36]
  FDI criteria for evaluation of restorations, percentage score.
  * Score: Properties
  * Clinically excellent/ very good: No secondary or primary caries.
  * Clinically good: Small and Localized 1. Demineralization, 2. Erosion or 3. Abfraction.
  * Clinically sufficient/satisfactory: Larger areas Of 1. Demineralization, 2. Erosion or 3. Abrasion/abfraction, dentine not exposed.
  * Clinically unsatisfactory: Caries with Cavitation and suspected undermining caries, 2. Erosion in dentine, 3.
  Abrasion/ abfraction in dentine.
  • Clinically poor: Deep caries or exposed dentine that is not accessible for repair of restoration.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Tezvergil-Mutluay, Professor, Study Chair — University of Turku
Locations (1):
- Horus University in Egypt, Damietta, Damietta Governorate, Egypt